CLINICAL TRIAL: NCT05082727
Title: Randomized, Double-blind, Placebo-controlled, Phase IIb Study, Safety Evaluation and Exploration of the Effect on Virologic Dynamics of Softgel KOVIR (TD.0068) in Combination With Background Therapy in Patients With Patients With COVID-19 Have Not Shown Signs of Acute Respiratory Failure.
Brief Title: Safety and Efficacy of Softgel KOVIR (TD0068) in the Combination Regimen With Background Treatment in COVID-19 Patients (KOVIR)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sao Thai Duong Joint Stock Company (Industry)
Collaborators: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOVIR-COVID19-2B
Record Dates: First submitted 2021-10-15; First posted 2021-10-19 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two arms: basic dose and placebo
Who Masked: Participant, Investigator
Masking Description: Double Blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KOVIR (TD0068) (Experimental): Standard dose, 5 capsules/time x 3 times/day x 14 days
  Interventions: Dietary Supplement: KOVIR (TD0068) oral softgel
- Placebo (Placebo Comparator): Placebo, 5 capsules/time x 3 times/day x 14 days
  Interventions: Dietary Supplement: Placebo oral softgel

INTERVENTIONS:
Dietary Supplement: KOVIR (TD0068) oral softgel — KOVIR (TD0068) is a softgel containing Allium sativum extract 270mg, Colostrum156.4 mg, fine powder mixed herbs 43.6mg
  Arms: KOVIR (TD0068)
Dietary Supplement: Placebo oral softgel — Placebo
  Arms: Placebo

SUMMARY:
The acute pneumonia pandemic caused by a new strain of corona virus 2019 named as COVID-19 by the World Health Organization (WHO) is a pandemic caused by SARS-CoV-2 virus. The reported symptoms vary from fever or chills, cough, shortness of breath, to muscle aches, headaches, loss of taste or smell.

The capsule KOVIR is a product based on the traditional medicine which is used to treat the cold conditions, also known as the initial plague according to the theory of traditional medicine.

DETAILED DESCRIPTION:
The acute pneumonia pandemic caused by a new strain of corona virus 2019 named as COVID-19 by the World Health Organization (WHO) is a pandemic caused by SARS-CoV-2 virus. The reported symptoms have included, but are not limited to fever or chills, cough, shortness of breath, muscle aches, headaches, loss of taste or smell, diarrhea, dizziness, sore throat, abdominal pain, anorexia, and vomiting.

The capsule KOVIR is a product based on the traditional prescription which is used to treat the cold conditions, also known as the initial plague according to the theory of traditional medicine.

The study timeline is expected from July 2021 to December 2022, including enrolment period, 14 days of treatment, data entry and analysis.

The study compares between standard dose regimen of KOVIR combined with background treatment in COVID-19 patients and placebo combined with background treatment in COVID-19 patients.

All participants will be treated and followed up in 14-day period. In case the participant meets the discharge criteria before 14 days, discontinuing the study drug will be done at the discretion of the investigators.

Screening procedures occur at Day 1. Periodic assessments are conducted daily from Day 2-14. Finally, End of study visit is conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age from 18 to 65 years old, Vietnamese nationality
* Participants diagnosed with Positive result of SARS-CoV-2 using real time RT-PCR test. - Quantitative test results for viral load > 4log and or CT value < 30 respiratory fluid samples with the time of sampling within 24 hours from the time of initiation of study treatment.
* Voluntary participation in the study by signing an informed consent
* Ability to adhere to treatment according to the investigator's assessment

Exclusion Criteria:

* Symptoms of severe influenza or severe acute respiratory infection (as defined by WHO).
* Acute reduction of ventilation function of respiratory apparatus and/or respiration function of the lung in any of the following three groups:

  * Respiratory distress due to hypoxemia with PaO2 less than 60mmHg when breathing room air.
  * Respiratory distress due to hypercapnia with PaCO2 above 50mmHg
  * Mixed respiratory distress accompanied by both a decrease in PaO2 and an increase in PaCO2
* Allergy/intolerance to any component of the study drug.
* Inability to administer medicine.
* Inability to comply with study procedures or to ensure compliance with study drug administration as assessed by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in viral load of SARS-CoV-2 | up to 14 days
  Daily assessment using qRT-PCR test
The time from baseline to the peak of viral load of SARS-CoV-2 | up to 14 days
  Daily assessment using qRT-PCR test
The time from baseline to no SARS-CoV-2 virus detection | up to 14 days
  Daily assessment using qRT-PCR test
Number of participants without SARS-CoV-2 virus detection after 7 days of treatment | after 7 days of treatment
  Assessment using qRT-PCR test
Number of participants without SARS-CoV-2 virus detection after 14 days of treatment | after 14 days of treatment
  Assessment using qRT-PCR test
Number of participants with respiratory distress complications requiring treatment | up to 14 days
  Appearance of symptoms of respiratory distress complications requiring treatment
Change in the severity of daily symptoms | up to 14 days
  Scale: 0 = Asymptomatic, 1 = Mild, 2 = Moderate, 3 = Severe
Number of Participants with Adverse Events as Assessed by CTCAE v5.0 | up to 30 days after last dose
  Study drug-related adverse events, adverse events leading to study termination, serious

CONTACTS AND LOCATIONS:
Overall Officials: Giang Tran, Dr.,MD., Principal Investigator — National hospital for tropical diseases
Locations (1):
- National hospital for tropical diseases, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: No